CLINICAL TRIAL: NCT04081883
Title: Decoding Islet Algorithms in Biosensors for Open and Closed-loop Glycemia Control in T1D Patients With Insulin Pump Coupled to Sensors.
Brief Title: Biosensors for Open and Closed-loop Glycemia Control in T1D Patients With Insulin Pump
Acronym: DIABLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2018/48
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Glucose Monitoring; Biosensor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biosensor algorithm (Experimental): The biosensor DIABLO algorithm is compared to Continuous Glucose Monitoring Systems (CGMS) utilisation.
  Interventions: Other: Biosensor algorithm

INTERVENTIONS:
Other: Biosensor algorithm — The biosensor DIABLO responses will be compared to the measurements of standard CGMS, using blood glucose measures every 10 minutes by taking interstitial fluid from Diabetes Type 1 (DT1) patients with an internal or external insulin pump.

SUMMARY:
In T1D, the destruction of beta-pancreatic cells causes insulin deficiency and requires insulin therapy whose control remains complex: even with recent technologies of continuous measurement and monitoring of blood glucose (CGM), current systems are electrochemical, insulin therapy algorithms do not are not optimal and cannot completely eliminate vital risks such as hypoglycemia. A new biosensor connected to the patient by microdialysis, will be tested in a clinical trial in CHU-Bdx on 10 T1D patients with an internal or external insulin pump. In various daily scenarios (meals, physical exercise) the biosensor DIABLO responses will be compared to the measurements of standard CGM systems.

DETAILED DESCRIPTION:
Continuous monitoring and linked drug delivery is a novel approach to the treatment of chronic diseases that provides powerful means to improve therapeutic outcomes and quality of patient's life. Type 1 diabetes (T1D) concerns 5 to 10% of the estimated 415 million cases of diabetes worldwide in 2016, expected to rise to 642 million by 2040(1). Continuous glucose monitoring systems (CGMS) linked to insulin delivery has provided a major advance(2). T1D is a serious, currently chronic and costly disease in children or young adults. Indeed, the destruction of pancreatic beta-cells leads to absolute insulin deficiency in T1D.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient with type 1 diabetes (T1D)
* Patient being equipped and trained with an external or internan insulin pump linked to a CGM
* Affiliated person or beneficiary of a social security scheme
* Free, informed and written consent

Exclusion Criteria:

* Patient under 18 years
* Patient not having T2D
* Pregnant or lactating patient
* No consent signed by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Comparison between biosensor to CGMS responses | 2 days after inclusion
  Measure blood glucose every 10 minutes by taking interstitial fluid from DT1 patients with an internal or external insulin pump to compare the biosensor responses to measurements of standard CGM systems.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan CATARGI, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Saint-André, Bordeaux, France